CLINICAL TRIAL: NCT01133587
Title: Patient Guided Psychiatric Admissions (Self-referral to Inpatient Beds)
Brief Title: Patient Guided Psychiatric Admissions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009/1704; 2009/1704 (Other Grant/Funding Number: St Olavs Hospital)
Record Dates: First submitted 2010-05-19; First posted 2010-05-31 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Schizophrenia; Bipolar Disorder
Keywords: Schizophrenia; bipolar disorder; Long term care; patient admission
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- admissions contract (Experimental): contract regarding "patient-guided admissions"
  Interventions: Behavioral: admissions contract
- wait list control (Active Comparator): 1 year on waiting list
  Interventions: Other: wait list control

INTERVENTIONS:
Other: wait list control — Patient-guided admissions contract regarding "patient-guided admissions" starting a year after.
  Arms: wait list control
Behavioral: admissions contract — contract regarding "patient-guided admissions" starting immediately
  Arms: admissions contract

SUMMARY:
To meet the requirement for increased patient involvement, several Community Mental Health Centres (CMHC) have initiated a service called "patient-guided admissions". The investigators will compare a group with "patient guided admission/self-referral to inpatient beds" with a group having treatment as usual.

It is expected that patients in the intervention group will experience more increased feeling of coping (patient activation) after 4 months and 12 months as a result of participating in "patient-guided admissions" than patients getting treatment as usual. In addition the total number of inpatient days either in the CMHC, psychiatric hospital or community rehabilitation centre is expected to be clearly lower in the intervention group than in the 'treatment-as-usual' group during one year after intake. Also the number of involuntary admissions either as inpatient or outpatient will be significant lower in the intervention group than the 'treatment-as-usual' group.The number of admissions in CMHC and psychiatric hospital, as well as the number of outpatient consultations in primary care, CMHC and psychiatric hospitals, will be lower in the intervention group than in the 'treatment-as-usual' group. Patients in the intervention group will experience improved mental health, increased feeling of coping (patient activation) and increased experience of recovery after 4 months and 12 months as a result of participating in "patient-guided admissions".

DETAILED DESCRIPTION:
Participants will be patients with psychosis or bipolar disorders. Patients in the intervention group will have a contract on "self-referral to inpatient beds" for one year. They can call the CMHC directly and ask for a bed for until 5 nights.

The patients in the 'treatment-as-usual' group will follow common procedures by either contacting their general practitioner, emergency department or duty doctor, and they will be offered a "self-referral to inpatient bed" contract after a year if they satisfy the inclusion criteria.

Regardless of the participation in the intervention group, the patients can also be ordinary admitted during the project period by a doctor via regular procedures in both hospital and CMHC if there is a need for this. All admissions will appear in the register data.

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia or bipolar disorder
* long term care
* established relationship with the ward

Exclusion Criteria:

* extensive substance use problems
* self-destructive behavior
* not able to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2010-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Patient activation/coping | 4 months
  Patient Activation Measure (PAM 13)
Patient activation/coping | 12 months
  Patient Activation Measure (PAM 13)

SECONDARY OUTCOMES:
Number of admissions | 12 months
  Number of admissions in CMHC, psychiatric hospital of community rehabilitation centre
Total number of inpatient days | 12 months
  Total number of inpatient days in CMHC, psychiatric hospital or community rehabilitation centre
Number of outpatient consultations | 12 months
  Number of outpatient consultations in primary care, in CMHC and psychiatric hospital
Number of involuntary admissions | 12 months
  Number of involuntary admissions either as inpatient or outpatient
Symptoms/functioning and recovery | 4 months
  Behavior and symptom identification scale (BASIS 32) and Recovery Assessment Scale (RAS 24)
Symptoms/functioning and recovery | 12 months
  Behavior and symptom identification scale (BASIS 32) and Recovery Assessment Scale (RAS 24)

CONTACTS AND LOCATIONS:
Overall Officials: Lasse Eriksen, PhD, Principal Investigator — St. Olavs Hospital
Locations (1):
- St.Olavs hospital, Psykisk helsevern, Nidaros DPS, Trondheim, Norway

REFERENCES:
- [Result] Moljord IE, Helland-Hansen KA, Salvesen O, Olso TM, Gudde CB, Rise MB, Steinsbekk A, Eriksen L. Short time effect of a self-referral to inpatient treatment for patients with severe mental disorders: a randomized controlled trial. BMC Health Serv Res. 2016 Sep 22;16(1):513. doi: 10.1186/s12913-016-1712-z. PMID 27659102
- [Result] Moljord IEO, Lara-Cabrera ML, Salvesen O, Rise MB, Bjorgen D, Antonsen DO, Olso TM, Evensen GH, Gudde CB, Linaker OM, Steinsbekk A, Eriksen L. Twelve months effect of self-referral to inpatient treatment on patient activation, recovery, symptoms and functioning: A randomized controlled study. Patient Educ Couns. 2017 Jun;100(6):1144-1152. doi: 10.1016/j.pec.2017.01.008. Epub 2017 Jan 11. PMID 28096034
- [Result] Sigrunarson V, Moljord IE, Steinsbekk A, Eriksen L, Morken G. A randomized controlled trial comparing self-referral to inpatient treatment and treatment as usual in patients with severe mental disorders. Nord J Psychiatry. 2017 Feb;71(2):120-125. doi: 10.1080/08039488.2016.1240231. Epub 2016 Oct 14. PMID 27739334